CLINICAL TRIAL: NCT06296355
Title: Impacts of Warning Labels on Ultra-Processed Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0300d
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Health Behavior; Diet, Healthy
Keywords: front-of-package labels; ultra-processed food; food and beverage purchases
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Warning Label (Experimental): Participants will view four products (a fruit-flavored drink, pretzels, a yogurt, and a breakfast cereal) each with a health warning label displayed on the front of package.
  Interventions: Behavioral: Health Warning Label
- Identity Warning Label (Experimental): Participants will view four products (a fruit-flavored drink, pretzels, a yogurt, and a breakfast cereal) each with an identity warning label displayed on the front of package.
  Interventions: Behavioral: Identity Warning Label
- Barcode Label (Other): Participants will view four products (a fruit-flavored drink, pretzels, a yogurt, and a breakfast cereal) each with a barcode control label displayed on the front of package.
  Interventions: Other: Barcode Label

INTERVENTIONS:
Behavioral: Health Warning Label — Message displayed on warning label is: "WARNING: Consuming ultra-processed food and drinks can cause weight gain, which increases the risk of obesity and type 2 diabetes."
  Arms: Health Warning Label
Behavioral: Identity Warning Label — Message displayed on warning label is: "WARNING: Ultra-processed food".
  Arms: Identity Warning Label
Other: Barcode Label — Barcode is displayed.
  Arms: Barcode Label

SUMMARY:
Purpose: The overall purpose of this study is to identify the impacts of an ultra-processed (UPF) health warning label and UPF identify warning label compared to a control label (i.e., a barcode).

Participants: ~4,000 US Latino adults of parental age (18-55 years), approximately 50% of whom will have limited English proficiency, recruited from a Latino-focused panel company.

Procedures: Participants will be randomly assigned to view food products with one of three label types: health warning labels, identity labels, or barcode control labels. Participants will be asked a series of questions about the products and the label they were assigned.

DETAILED DESCRIPTION:
On the study platform (Qualtrics), participants will be randomly assigned to 1 of 3 arms with equal probability: a UPF health warning label, a UPF identity label, or a barcode control label. Participants will view four products (a fruit-flavored drink, pretzels, a yogurt, and a breakfast cereal) displayed in random order, each with a label displayed on the front of package according to the participants' study arm. Participants will complete a 13-item online survey to assess each product as to a) whether the product is ultra-processed; b) perceptions of healthfulness; c) intentions to purchase the product.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as Latino or Hispanic
* Ages 18-55 years old
* Currently resides in the United States

Exclusion Criteria:

* Not identifying as Latino or Hispanic
* Less than 18 or greater than 55 years old
* Not residing in the United States

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4000 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Identification of a product as ultra-processed | Immediately after exposure to intervention, assessed during 1-time online study visit.
  Correct identification of a product as ultra-processed. Measured with the question, "Do you think this product is ultra-processed?" Response options are Yes, No, and I'm not sure.

SECONDARY OUTCOMES:
Perceived product healthfulness of ultra-processed products | Immediately after exposure to intervention, assessed during 1-time online study visit.
  Measured with the question, "How good or bad for your health would it be to consume this product every day?" Likert responses are on a 1 to 5 scale, from "Very bad" (coded as 1) to "Very good" (coded as 5), with higher scores representing a higher perceived healthfulness.
Intentions to purchase ultra-processed products | Immediately after exposure to intervention, assessed during 1-time online study visit.
  Measured with the question, "How likely would you be to purchase this product in the next week, if it were available?" Likert responses are on a 1 to 5 scale, from "Not at all likely" (coded as 1) to "Extremely likely" (coded as 5), with higher scores representing a higher intention to purchase ultra-processed products.
Perceived message effectiveness | Immediately after exposure to intervention, assessed during 1-time online study visit.
  Measured with the question, "How much does this message discourage you from wanting to consume an ultra-processed food or drink?" Likert responses are on a 1 to 5 scale, from "Not at all" (coded as 1) to "Very much" (coded as 5), with higher scores representing a higher perceived message effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Smith Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Carolina Population Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset and the corresponding survey codebook will be shared beginning 9 months and continuing for 36 months after publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC. The study protocol, statistical analysis plan, and informed consent form will be published alongside as supplementary material.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 36 months following publication of study results.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT06296355/SAP_000.pdf